CLINICAL TRIAL: NCT05346757
Title: Prospective, Multicenter, Comparative, Paired Study to Validate a microRNA-based Fecal Test for Colorectal Cancer Screening. The miRFec Study
Brief Title: Validation of a microRNA-based Fecal (miRFec) Test for Colorectal Cancer Screening, Surveillance and Diagnosis
Acronym: miRFec
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Antoni Castells, Principal investigator, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: miRFec001
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Once the participant accepts to participate in the study, a fecal sample collection kit will be delivered together with the sample collection instructions. The sample must be collected at home before starting bowel preparation, more specifically between 24-72 hours before the day that colonoscopy is scheduled. Both miRNA expression and FIT will be analyzed in a central laboratory (Hospital Clinic of Barcelona) from the same fecal sample.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- miRFec test (Other): The miRFec test corresponds to the combination of fecal hemoglobin concentration and fecal miRNA expression
  Interventions: Diagnostic Test: miRFec test

INTERVENTIONS:
Diagnostic Test: miRFec test — The miRFec test actually corresponds to the combination of fecal hemoglobin concentration (ie. FIT) and fecal miRNA expression

SUMMARY:
The present study aims to compare effectiveness and cost-effectiveness of the miRFec test with respect to fecal immunochemical test (FIT) for the detection of advanced colorectal neoplasm among individuals participating in colorectal cancer (CRC) screening, surveillance and diagnosis.

DETAILED DESCRIPTION:
The miRFec test -a Gradient Boosting Machine-generated algorithm that includes two fecal miRNAs (miR-421 and miR-27a-3p) and fecal hemoglobin concentration, along with age and gender- is more effective and cost-effective than FIT for the identification of patients with advanced colorectal neoplasm (i.e. colorectal cancer, advanced adenomas or advanced serrated lesions) among individuals participating in colorectal cancer screening and surveillance programs, and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 50 to 75 (average-risk) referred to colonoscopy-based CRC screening.
* Male or female aged 30 to 80 with family history of CRC (moderate-risk) referred to colonoscopy-based CRC screening.
* Male and female aged 18 or older with personal history of colorectal polyps referred to colonoscopy surveillance.
* Male and female aged 18 or older with personal history of CRC referred to colonoscopy surveillance.
* Male and female aged 18 or older with colorectal symptoms referred to diagnostic colonoscopy.

Exclusion Criteria:

* Lack of informed consent to participate
* Personal history of Lynch syndrome
* Personal history of adenomatous or hamartomatous polyposis
* Personal history of serrated polyposis syndrome
* Personal history of inflammatory bowel disease
* Personal history of total colectomy for any reason
* Family history of Lynch syndrome
* Family history of adenomatous or hamartomatous polyposis
* Family history of serrated polyposis syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5390 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for advanced colorectal neoplasm | Through study completion, an average of 3 years
  To compare the sensitivity of the miRFec test with respect to FIT for the detection of advanced colorectal neoplasm

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 3 years
  To compare the specificity of the miRFec test with respect to FIT
Sensitivity for colorectal cancer | Through study completion, an average of 3 years
  To compare the sensitivity of the miRFec test with respect to FIT for the detection of colorectal cancer
Sensitivity for advanced adenomas | Through study completion, an average of 3 years
  To compare the sensitivity of the miRFec test with respect to FIT for the detection of advanced adenomas
Sensitivity for advanced serrated lesions | Through study completion, an average of 3 years
  To compare the sensitivity of the miRFec test with respect to FIT for the detection of advanced serrated lesions
Detection rate for advanced colorectal neoplasm | Through study completion, an average of 3 years
  To compare the detection rate for advanced colorectal neoplasm of the miRFec test with respect to FIT
Discrimination capacity for advanced colorectal neoplasms | Through study completion, an average of 3 years
  To compare the discrimination capacity of the miRFec score and fecal hemoglobin concentration for the detection of advanced colorectal neoplasm
Discrimination capacity for colorectal cancer | Through study completion, an average of 3 years
  To compare the discrimination capacity of the miRFec score and fecal hemoglobin concentration for the detection of colorectal cancer
Cost-effectiveness for advanced colorectal neoplasm detection | Through study completion, an average of 3 years
  To compare the cost (euros) for detecting one advanced colorectal neoplasm using the miRFec test with respect to the corresponding figure using FIT

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Castells, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After the end of the study
Access Criteria: Request to the study's principal investigator

REFERENCES:
- [Background] Duran-Sanchon S, Moreno L, Auge JM, Serra-Burriel M, Cuatrecasas M, Moreira L, Martin A, Serradesanferm A, Pozo A, Costa R, Lacy A, Pellise M, Lozano JJ, Gironella M, Castells A. Identification and Validation of MicroRNA Profiles in Fecal Samples for Detection of Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):947-957.e4. doi: 10.1053/j.gastro.2019.10.005. Epub 2019 Oct 14. PMID 31622624
- [Result] Duran-Sanchon S, Moreno L, Gomez-Matas J, Auge JM, Serra-Burriel M, Cuatrecasas M, Moreira L, Serradesanferm A, Pozo A, Grau J, Pellise M, Gironella M, Castells A. Fecal MicroRNA-Based Algorithm Increases Effectiveness of Fecal Immunochemical Test-Based Screening for Colorectal Cancer. Clin Gastroenterol Hepatol. 2021 Feb;19(2):323-330.e1. doi: 10.1016/j.cgh.2020.02.043. Epub 2020 Feb 28. PMID 32113893

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05346757/Prot_SAP_ICF_002.pdf